CLINICAL TRIAL: NCT02254096
Title: Safety, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BIRT 1696 BS as a Solution (10, 100, 400, 1000, 2000, 3000 mg) in 15 ml PEG 400 to Healthy Human Subjects. A Three Part Study: Part 1 Placebo-controlled, Randomised, Dose Escalating Double Blinded Within Each Dose Level; Part 2 Open Label Grapefruit Juice Effect in 100 mg Dose Level Group; Part 3 Open Label Food Effect in 400 mg Dose Level Group
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of BIRT 1696 BS in Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1195.1
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (4):
- BIRT 1696 BS (Experimental): single escalating dose phase
  Interventions: Drug: BIRT 1696 BS
- BIRT 1696 BS + GFJ (Experimental): single dose grapefruit effect arm
  Interventions: Drug: BIRT 1696 BS; Other: Grapefruit juice (GFJ)
- BIRT 1696 BS + HFM (Experimental): single dose food effect arm
  Interventions: Drug: BIRT 1696 BS; Other: High fat meal (HFM)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIRT 1696 BS
  Arms: BIRT 1696 BS; BIRT 1696 BS + GFJ; BIRT 1696 BS + HFM
Drug: Placebo
  Arms: Placebo
Other: Grapefruit juice (GFJ)
  Arms: BIRT 1696 BS + GFJ
Other: High fat meal (HFM)
  Arms: BIRT 1696 BS + HFM

SUMMARY:
The objectives are:

1. To assess safety, pharmacokinetics, and pharmacodynamics of BIRT 1696 BS in rising single doses.
2. To assess safety, pharmacokinetics, and pharmacodynamics of single dose of 100 mg BIRT 1696 BS after grapefruit juice.
3. To asses safety and pharmacokinetics of single dose of 400 mg BIRT 1696 BS after a 67 g fat and high caloric breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age ≥18 and ≤60 years
* Body Mass Index ≥18.5 and ≤29.9 kg/m2

Exclusion Criteria:

* Female subjects who are lactating or of child bearing potential as defined by surgically sterile or post menopausal (no periods for at least 12 months and elevated follicle stimulating hormone with low estradiol while on no estrogen supplementation unless surgically sterile). Females should use barrier contraception (e.g. condoms) prior to administration of study medication, during the study and at least one month after release from the study. Women must have had negative blood pregnancy tests
* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial, (< 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (< 2 months prior to administration or during trial)
* Smoker (> 10 cigarettes or >3 cigars or >3 pipes/day)
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Use of methylxanthine-containing drinks or foods (coffee, tea, cola, energy drinks, chocolate, etc.), grapefruit or grapefruit juice, alcohol, green tea, or tobacco < 5 days prior to administration of study drug or during trial
* Blood donation or loss > 400 mL, < 1 month prior to administration or during the trial
* Excessive physical activities < 5 days prior to administration of study drug or during trial
* Clinically relevant laboratory abnormalities
* Any ECG value outside of the reference range of clinical relevance including, but not limited to QRS interval > 110 ms or QTcB > 450 ms (males) or QTcB > 470 ms (females)
* Inability to comply with dietary regimen of study centre
* Inability to comply with the investigator's instructions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2002-05; Primary Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 44 days
Number of subjects with clinically significant changes in vital signs | up to 44 days
Number of subjects with abnormal changes in laboratory parameters | up to 44 days
Number of subjects with abnormal findings in electrocardiogram | up to 44 days
Number of subjects with abnormal findings in physical examination | up to 44 days
Assessment of tolerability on a verbal rating scale | up to 44 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | up to 48 hours after drug administration
Total area under the plasma drug concentration-time curve from time zero to infinity (AUC0-∞) | up to 48 hours after drug administration
Time to the maximum plasma concentration (tmax) | up to 48 hours after drug administration
Elimination half-life (t1/2) | up to 48 hours after drug administration
Total apparent oral clearance of drug from plasma after oral administration (CL/F) | up to 48 hours after drug administration
Apparent volume of distribution based on terminal elimination phase, divided by F (bioavailability factor) (Vz/F) | up to 48 hours after drug administration
Mean residence time (MRT) | up to 48 hours after drug administration
Urinary excretion | up to 24 hours after drug administration
Receptor occupancy as determined by binding of anti-lymphocyte function associated antigen-1 antibody fragment (Fab) | up to 168 hours after drug administration
Inhibition of superantigen induced interleukin-2 production ex vivo | up to 168 hours after drug administration